CLINICAL TRIAL: NCT06734975
Title: Effect of Intraoperative Superior Laryngeal Nerve Blocks on Patient Outcomes in Microdirect Laryngoscopy for Benign Vocal Fold Lesions: A Randomized Trial
Brief Title: Effect of Superior Laryngeal Nerve Blocks on Patient Outcomes in Laryngeal Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Kenneth Yan, MD, PhD, Assistant Professor, Laryngology, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2024002226
Record Dates: First submitted 2024-12-03; First posted 2024-12-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Vocal Cord Disease; Vocal Cord Polyp; Vocal Cord Cyst
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Superior laryngeal nerve block (Experimental): Patients will receive a superior laryngeal nerve block consisting of 1 milliliter of 0.25% bupivacaine and milliliter of triamcinolone acetate 40 mg/ml to the neck on the side of the vocal cord lesion during their surgery.
  Interventions: Drug: Superior laryngeal nerve block - Intervention (Bupivacaine and triamcinolone acetonide suspension)
- Placebo (Placebo Comparator): Patients will receive a placebo of 2 milliliter saline injection to the neck on the side of the vocal cord lesion during their surgery.
  Interventions: Drug: Superior laryngeal nerve block - Placebo (saline)

INTERVENTIONS:
Drug: Superior laryngeal nerve block - Intervention (Bupivacaine and triamcinolone acetonide suspension) — Patients will receive a superior laryngeal nerve block consisting of 1 ml of 0.25% bupivacaine and 1mL of triamcinolone acetate 40 mg/ml to the neck on the side of the vocal cord lesion during their surgery.
  Arms: Superior laryngeal nerve block
Drug: Superior laryngeal nerve block - Placebo (saline) — Patients will receive a saline placebo of 2mL saline to the neck on the side of the vocal cord lesion during their surgery.
  Arms: Placebo

SUMMARY:
Patients undergoing surgery on their vocal cord will either receive a numbing injection to their throat or a saline injection during surgery. Symptoms such as how much coughing or pain patients have after surgery, as well as whether patient's voice gets better will be interrogated.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 18 years or older at time of consent
* Patient has suspected or confirmed benign vocal fold lesion
* Patient is planning to undergo direct laryngoscopy with excision of the vocal fold lesion
* Patient is English or Spanish speaking
* Patient is not pregnant per self report
* Patient is not incarcerated

Exclusion Criteria:

* Patient is not 18 years of age or older at consent date
* Patient does not speak English or Spanish
* Patient is currently pregnant or plans to become pregnant prior to their study procedure
* Patient has a laryngeal malignancy or found to find a laryngeal malignancy on final pathology
* Patient will not be undergoing direct laryngoscopy with excision of lesion
* Patient is unable to provide consent or complete study activities
* Patient is incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 1, 3 and 7 days after surgery
  We will record postoperative pain via the 100 mm visual analog scale (VAS). The minimum is 0, maximum is 100, and a higher score indicates more pain and thus a worse outcome.
Postoperative cough | Follow up appointment 2-4 weeks after surgery
  Cough severity index score. The Cough Severity Index (CSI) is a validated 10 question survey about cough severity with each question rated on a Likert Scale from 0-4, where 4 is most severe. The maximum score is 40 and the minimum score is 0, where 40 represents the most severe cough.
Postoperative voice outcome | Postoperative appointment 2-4 weeks after surgery
  Voice Handicap Index-10 (VHI-10) score. The VHI-10 is a validated 10 question survey about quality of life related to dysphonia with each question rated on a Likert Scale from 0-4, where 4 is most severe. The maximum score is 40 and the minimum score is 0, where 40 represents the most vocal handicap.

SECONDARY OUTCOMES:
Post-extubation cough | 5 minutes postoperative
  Clinical assessment of cough immediately following extubation from surgery using the following scale:
  * Grade 0: No cough.
  * Grade 1: Mild cough - the patient has occasional coughing that does not interfere with recovery or cause noticeable discomfort. No intervention is required.
  * Grade 2: Moderate cough - more than 1 episode of unsustained coughing lasting over 64 seconds causing discomfort and may temporarily delay recovery. Requires minimal supportive interventions (hydration, suctioning).
  * Grade 3: Severe cough - intense or continuous coughing lasting over 64 seconds that causes significant discomfort, delays recovery, or contributes to complications such as wound dehiscence or an airway obstruction. May require a medical intervention such as nebulization or repositioning.
  Grade 3 represents the worst outcome, characterized by significant discomfort, delayed recovery, or complications requiring medical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Yan, MD, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers New Jersey Medical School, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No